CLINICAL TRIAL: NCT03762889
Title: Peri-operative Application of EYEPROTX General Anesthesia Protective Goggles as an Effective Modality to Reduce the Incidence of Corneal Injury Post-Intubation.
Brief Title: Peri-operative Application of Eyeprotx General Anesthesia Goggles As Prevention Against Corneal Injury Post Intubation.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial no longer occurring.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Leo Kleyman, Research Fellow, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180875
Record Dates: First submitted 2018-11-20; First posted 2018-12-04 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Corneal Injuries
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Intervention Model Description: In this cohort study, 100 preoperative patients from Jackson Memorial Hospital would be randomly assigned based on age, gender, and type of anesthesia to three samples: anesthesia with Eyeprotx™ Goggles, anesthesia with eyelid tape, and anesthesia with ointment application. Analysis of samples will be based on length of procedure, length of preventative measure application, position during operation(supine or prone), and postoperative events. Patient discomfort or pain, eye dryness intensity would be rated on numerical rating scale. Qualitative analysis will include additional comments from patients and the anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Eyeprotx™ Group (Experimental): This group of participants will use the Eyeprotx™ General Anesthesia Protective Goggles when intubated perioperatively under general anesthesia.
  Interventions: Device: Eyeprotx™ General Anesthesia Protective Goggles
- Eyelid Tape Group (Active Comparator): This group of participants will be receiving the eyelid tape as the preventative measure when intubated perioperatively under general anesthesia.
  Interventions: Device: Eyelid Tape
- Eye Ointment Group (Active Comparator): This group of participants will be receiving the ointment application when intubated perioperatively under general anesthesia.
  Interventions: Device: Eye Ointment

INTERVENTIONS:
Device: Eyeprotx™ General Anesthesia Protective Goggles — Eyeprotx™ Protective Goggles have been designed specifically for use in the operating room or in any scenario where general anesthesia must be used, such as intubation in an emergency. The integral function is to reduce intraocular pressure while in place, prevent operating room bright light penetration, facilitate a swift placement preventative measure with straps, form a barrier against bacterial invasion and mechanical damage. This study would seek to examine this goggles' effectiveness as a preventative measure as vs. other measures.
  Arms: Eyeprotx™ Group
Device: Eyelid Tape — Taping the eyelids during intubation is one of the standard techniques used perioperatively under general anesthesia. This intervention would be used for the Eyelid Tape Group.
  Arms: Eyelid Tape Group
Device: Eye Ointment — Another standard technique used perioperatively under general anesthesia is to apply an ointment to the eye for lubrication. This intervention would be applied to the Eye Ointment Group.
  Arms: Eye Ointment Group

SUMMARY:
This is a randomized controlled trial that seeks to examine the effectiveness of Eyeprotx™ protective goggles in comparison to traditional methods against ocular injury that can occur perioperatively under general anesthesia.

DETAILED DESCRIPTION:
Ocular injury is but a devastating condition that can occur perioperatively under general anesthesia. Corneal abrasion is the most common ocular injury during general anesthesia, surpassing case incidence of damage caused by patient movement in ophthalmologic surgery. Causes of ocular injury include corneal drying due to the suppression of tear ducts from anesthetic agents, direct physical trauma, or agitation from the volatile anesthetic used. Ocular injury may also occur due to bacterial infection with MRSA, preventative methods, or rubbing of the eyes postoperatively due to agitation. Agitation may be caused by corneal drying or by shift or disruption in rapid eye movement sleep cycle from light penetration through the eyelids. Attempts at prevention of corneal abrasion have been used, including taping the eyelids shut, manual eye closure, paraffin-based ointment application into the conjunctival sac, and the use of hydrophilic contact lenses, although only a few studies have validated the comparison of these methods' effectiveness.

Eyeprotx™ Protective Goggles have been designed specifically for use in the operating room or in any scenario where general anesthesia must be used, such as intubation in an emergency. Current ocular protective measures such as tapes during anesthesia have been associated with injury and infection. With this study, we hope to find a safer preventative technique against ocular injury during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia
* Patients admitted to Jackson Memorial Hospital

Exclusion Criteria:

* Patients unable to communicate, for whatever reason
* Patients predisposed to eye conditions
* Patients with history of increased intraocular pressure
* Patients with a medical history of Sicca syndrome
* Patients with claustrophobia
* Patients with pseudoexfoliation syndromes
* Patients with a current exopthalmic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Baseline Ocular Condition post-operatively | The patient's initial rating will be recorded approximately ten minutes before surgery at the point of anesthesia evaluation and will be reassessed up to 24 hours post-operatively.
  The following will be measured upon evaluation, using a numerical scale of 1 to 8, with 1 being complete absence of condition and 8 being the most severe presentation of the condition:
  1. eye discomfort, 2, pain, and 3. dryness intensity, each on a numerical rating-scale of 1 to 8, The measures will be compared among the goggle, ointment, and tape groups.
Incidence of Ocular Complications post-operation | Evaluation of these complications will be done from the point the patient has returned to the recovery room to up to one week post-surgery or until discharge, whichever comes first.
  Incidence of corneal abrasion, conjunctivitis, MRSA infection, and direct ocular trauma will be assessed by the anesthesiologist or nurse anesthetist and will be recorded upon diagnosis of condition for all groups.

SECONDARY OUTCOMES:
Patient Awareness during Anesthesia | This measure will be evaluated up to 48 hours post-surgical operation.
  Patient awareness of being under anesthesia will be recorded qualitatively, with accounts of anxiety and/or fear being noted, if applicable.
Incidence of Nightmare during Use | This measure will be evaluated up to 48 hours post-surgical operation.
  Patient's report of experiencing nightmares during the surgery will be recorded qualitatively.

OTHER OUTCOMES:
Usability Scale Per Operator | This measure will be evaluated up to 6 months after the post-surgical operation.
  The anesthesiologists and nurse anesthetists working on the trial will be asked to complete a usability scale questionnaire to evaluate the effectiveness of the different variation of the goggles, such as goggles with a strap versus goggles with short sterilized adhesive tape.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Au, DO MD PHD, Principal Investigator — Jackson Health System
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gild WM, Posner KL, Caplan RA, Cheney FW. Eye injuries associated with anesthesia. A closed claims analysis. Anesthesiology. 1992 Feb;76(2):204-8. doi: 10.1097/00000542-199202000-00008. PMID 1736697
- [Background] Figueiro MG, Rea MS. Preliminary evidence that light through the eyelids can suppress melatonin and phase shift dim light melatonin onset. BMC Res Notes. 2012 May 7;5:221. doi: 10.1186/1756-0500-5-221. PMID 22564396
- [Background] White E, Crosse MM. The aetiology and prevention of peri-operative corneal abrasions. Anaesthesia. 1998 Feb;53(2):157-61. doi: 10.1046/j.1365-2044.1998.00269.x. PMID 9534639
- See also: "Corneal Injuries During General Anesthesia", Snow et al — https://journals.lww.com/anesthesia-analgesia/Abstract/1975/07000/Corneal_Injuries_During_General_Anesthesia.14.aspx